CLINICAL TRIAL: NCT01081561
Title: Randomized Study of Corneal Collagen Cross-Linking With the UV-X System for the Treatment of Keratectasia in Eyes With Intacs Compared to Eyes Without Intacs
Brief Title: Collagen Cross-Linking for Keratoconus/Ectasia With and Without Intacs
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yaron S. Rabinowitz M.D. (Other)
Responsible Party: Sponsor-Investigator, Yaron S. Rabinowitz M.D., Yaron S Rabinowitz M.D., Cornea Genetic Eye Institute
Organization: Cornea Genetic Eye Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #20090780
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2017-12

CONDITIONS: Keratoconus; Ectasia
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cross-linking (Active Comparator): Corneal collagen cross-linking with riboflavin and UVA light
  Interventions: Drug: Riboflavin
- Cross-linking plus INTACS (Active Comparator): Corneal collagen cross-linking with riboflavin and UVA light plus INTACS
  Interventions: Drug: Riboflavin

INTERVENTIONS:
Drug: Riboflavin — Removal of the epithelium, riboflavin drops every 2 minutes for 30 minutes follow by UV light radiation and addition riboflavin drops every 2 minutes for 30 minutes. Some subjects will be randomized to recieve INTACS prior to treatment with riboflavin.
  Other Names: Peschke Meditrade

SUMMARY:
This study will determine the efficacy of collagen cross linking for progressive keratoconus and ectasia after lasik. It will try and determine which is a more effective treatment: collagen cross linking alone or collagen cross linking combined with Intacs, a treatment which has already been proven to be effective in decreasing corneal curvature in patients with keratoconus.

DETAILED DESCRIPTION:
In this study we will attempt to determine whether Collagen Cross Linking alone, one combined with insertion of INTACS is the most effective treatment for patients with progressive keratoconus in patients who have progressive disease.

These treatments have been widely used outside of the United States for the treatment of progressive keratoconus. Corneal Collagen Cross linking was recently approved in the United States for the treatment of progressive keratoconus. We will attempt to study 600 patients total. 300 patients will be assigned to cross linking only while another 300 will be assigned to cross linking and INTACS. Once adequate number of study subjects have been recruited data will be analyzed to determine which treatment is more effective. The following parameters from Topography, OCT and Tomography will be studied(these are Max K(pentacam) Kvalue(Tomey Topography)I-Svalue(Tomey Topography Astigmatism(Tomey Topography) and Min OCT(corneal pachymetry) any one of these metrics that achieve a value of 1 or more will be included in the analysis since the cornea is so irregular that values less than one could be artifact

ELIGIBILITY:
Inclusion Criteria:

* progressive keratoconus or ectasia

Exclusion Criteria:

* cornea thinner than 400um
* K readings greater than 60D
* Central corneal scarring

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2009-01-21 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of UV-X cross linking to halt progression of keratoconus | 10 years
  Any change of 1 or more of the following indices will be classified as progression. The following parameters will be studied Max K, Steep K, I-S value,Min OCT(pachymetry

CONTACTS AND LOCATIONS:
Overall Officials: Yaron S Rabinowitz, M.D., Principal Investigator — Cornea Genetic Eye Institute; Ezra Maguen, M.D., Principal Investigator — american eye institute; Yuri Oleynikov, M.D. PhD, Principal Investigator — Cornea Genetic Eye Institute; James Salz, M.D., Principal Investigator — Laser Eye Associates; Ronald Gaster, MD, Principal Investigator — Cornea Eye Institute, Beverly Hills
Locations (1):
- Cornea Eye Institute, 50 North La Cienaga Blvd, #340, Beverly Hills, California, United States

IPD SHARING:
Plan to Share IPD: No